CLINICAL TRIAL: NCT07102472
Title: Community Immunity Versus Herd Immunity
Brief Title: An Experiment Comparing Public Reactions to the Labels "Community Immunity" Versus "Herd Immunity".
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: commimm
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Attitudes
MeSH Terms: conditions — Behavior | interventions — Immunity, Herd

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herd immunity (Placebo Comparator)
  Interventions: Behavioral: Herd immunity
- Community immunity (Experimental)
  Interventions: Behavioral: Using the term "community immunity" instead of "herd immunity"

INTERVENTIONS:
Behavioral: Using the term "community immunity" instead of "herd immunity" — In the intervention arm, participants are shown the less traditional term "community immunity" in place of the more traditional "herd immunity"
  Arms: Community immunity
Behavioral: Herd immunity — Using the traditional term "herd immunity"
  Arms: Herd immunity

SUMMARY:
Participants are shown a scenario consisting of static images from a previous study ("herdimm") showing a visualization of how herd immunity works. Participants are randomized to see the text with the term "herd immunity" or "community immunity."

ELIGIBILITY:
Inclusion Criteria:

* Able to use a computer
* Able to use the internet
* Able to read and respond to questions in English or French
* 18+ years old and living in Canada

Exclusion Criteria:

- Unable to view images on a computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-07-22 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Orientation towards protection of others | Immediately after the intervention
  A measure of the extent to which people believe that individual vaccination behavior is important to protect others. Question wording: "When a safe and effective vaccine exists that can prevent people from catching and passing on a contagious disease, it is important for people to get vaccinated to protect ..." Measured across two to three items (family, others in the community, people who are more vulnerable to disease) on a 7-point Likert-type scale (strongly disagree = 1, strongly agree = 7).

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be deposited on Borealis, Laval University's official data repository.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD and supporting information will be available when the study report is complete.
Access Criteria: Anyone with internet access will be able to access the public-facing file. Some data may require access through Borealis registration.
URL: https://borealisdata.ca/